CLINICAL TRIAL: NCT04408092
Title: Pilot Study of the Effect of GM-CSF on Macrophages in Incompletely Resected or Recurrent Ependymoma
Brief Title: Study of the Effect of GM-CSF on Macrophages in Ependymoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0133.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2020-05-29 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ependymoma, Recurrent Childhood; Ependymoma
Keywords: granulocyte macrophage colony stimulation factor; Incomplete resection
MeSH Terms: conditions — Ependymoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: standard treatment of EPN includes repeat surgeries at (1) second-look surgery to remove residual tumor after first-look surgery at initial diagnosis, and (2) optimal debulking of recurrent tumor, providing a rare opportunity to measure the effect of experimental therapy directly in children's brain tumors. Ten patients each will be entered into the second-look and recurrence strata of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GM-CSF treatment at second-look surgery arm (Experimental): Newly diagnosed patients with EPN who have a subtotal resection at initial presentation and are without evidence of metastatic tumor will be enrolled in this stratum. Total patient population in this stratum will be 10 patients. It should be noted that prior experience suggests that about 1/3 of newly presenting patients still have residual tumor after the initial surgery
  Interventions: Drug: Granulocyte Macrophage Colony Stimulation Factor
- GM-CSF treatment at recurrence arm. (Experimental): EPN patients with a first regional relapse and without evidence of metastatic tumor will be enrolled in this stratum. Total patient population will be 10 patients.
  Patients with a first recurrence will have the recurrence confirmed by the local institutional neuro-radiologists. They will have the entire neuro-axis scanned and a spinal tap performed (where safe) to exclude metastatic tumor. They will then receive 5 days of GM-CSF and then proceed to surgery if deemed clinically indicated by the treating physician
  Interventions: Drug: Granulocyte Macrophage Colony Stimulation Factor

INTERVENTIONS:
Drug: Granulocyte Macrophage Colony Stimulation Factor — Recombinant Granulocyte Macrophage Colony Stimulation Factor (rGM-CSF) is a hematopoietic growth factor which supports survival, clonal expansion, and differentiation of hematopoietic progenitor cells. rGM-CSF induces partially committed progenitor cells to divide and differentiate in the granulocyte-macrophage pathways. rGM-CSF stimulates the production of monocytes, granulocytes, erythrocytes, and sometimes, megakaryocytes in the bone marrow. It also induces mature macrophages to increase phagocytosis, superoxide generation, Antibody Dependent Cell-mediated Cytotoxicity (ADCC), tumoricidal killing and cytokine production (IL-1 and tumor necrosis factor). GM-CSF was used in the first successful phase III trial of immunotherapy in the pediatric COG protocol, ANBL0931, a national study in high risk neuroblastoma.
  Other Names: GM-CSF

SUMMARY:
This study plans to learn more about the use of Granulocyte Macrophage Colony Stimulation Factor (GM-CSF) on ependymoma tumors. The use of GM-CSF is a potential way of increasing the infiltration of immune cells and this study is looking at whether or not this will improve the outcome of patients with an ependymoma

DETAILED DESCRIPTION:
To study whether Granulocyte Macrophage Colony Stimulation Factor (GM-CSF) increases macrophage infiltration in children with ependymoma (EPN) who are to have planned surgery as a standard procedure for incomplete resection or recurrent tumor. To correlate the extent of macrophage infiltration with other immune markers of the tumor at subsequent surgery with outcome. This is intended as a pilot protocol with the potential to be incorporated in the next COG (Children's Oncology Group) national ependymoma studies.

Recombinant Granulocyte Macrophage Colony Stimulation Factor (rGM-CSF) is a hematopoietic growth factor which supports survival, clonal expansion, and differentiation of hematopoietic progenitor cells. rGM-CSF induces partially committed progenitor cells to divide and differentiate in the granulocyte-macrophage pathways. rGM-CSF stimulates the production of monocytes, granulocytes, erythrocytes, and sometimes, megakaryocytes in the bone marrow. It also induces mature macrophages to increase phagocytosis, superoxide generation, Antibody Dependent Cell-mediated Cytotoxicity (ADCC), tumoricidal killing and cytokine production (IL-1 and tumor necrosis factor).

Registration of all participants must occur before any study-related procedures. Staff will be available to register participants Monday thru Friday, from 8:00 AM to 5:00 PM Mountain Standard Time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 months and < 21 years at the time of study enrollment.
* Patients must be one of the following:

  • Newly diagnosed with posterior fossa ependymoma with a subtotal resection at initial surgery. These patients will be eligible for stratum 1.
  * Be in first relapse of their posterior fossa ependymoma. These patients will be eligible for stratum 2.
* Histologically confirmed diagnosis of intracranial ependymoma .
* Pre or post-operative MR imaging of the brain demonstrates no evidence of non-contiguous spread beyond the primary site
* Pre or post-operative MR imaging of the spine demonstrates no evidence of non-contiguous spread beyond the primary site
* Pre-operative CSF cytology obtained from the lumbar CSF space demonstrated no evidence of non-contiguous spread beyond the primary site.

  • The requirement for lumbar CSF examination may be waived if deemed to be medically contraindicated.
* Patients must meet one of the following performance scores.

  • ECOG performance status scores of 0, 1, or 2.
  * Karnofsky score of ≥ 50 for patients > 16 years of age or Lansky score of ≥ 50 for patients ≤ 16 years of age
* Organ Function Requirements:

Adequate renal function defined as:

* Creatinine clearance or radioisotope GFR ³ 70ml/min/1.73 m2 or
* A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female

1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5

1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

* Adequate liver function defined as:
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
* SGOT (AST) or SGPT (ALT) < 3 x upper limit of normal (ULN) for age.
* Patients with Gilbert syndrome or hemolytic anemia are eligible if total bilirubin is < 3 x upper limit of normal (ULN) for age.
* Adequate Bone Marrow Function defined as:
* Peripheral absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count >= 100,000/uL (transfusion independent).

Exclusion Criteria:

* Patients with a diagnosis of spinal cord ependymoma, myxopapillary ependymoma, subependymoma, ependymoblastoma, supratentorial ependymoma, or mixed glioma are NOT eligible.
* Patients with evidence of metastatic disease by MRI or CSF cytology are NOT eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with increased M/M infiltration compared to institutional and ACNS0121 controls | 8 years
  Outcome measure is met if cell count is >50 AIF1+ microglia per high power field (40x)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Foreman, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Denver, Colorado
  - Arnold Palmer Hospital for Children, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No